CLINICAL TRIAL: NCT03055819
Title: Evaluation of Patient and Physician Satisfaction With the Zift eLevatIon of Facial Tissue Clinical Study
Acronym: LIFT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company no longer exists
Sponsor: Zift, LLC (Industry)
Collaborators: Libra Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1068-001Rev3
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Senile Ptosis
Keywords: Brow Lift; Brow Ptosis

STUDY DESIGN:
Intervention Model Description: Single arm, open label, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ZiftLift Tissue Anchor (Experimental): Use of ZiftLift Tissue Anchors for Brow Lift
  Interventions: Device: Brow Lift

INTERVENTIONS:
Device: Brow Lift — Minimally Invasive Brow Lift
  Other Names: Brow Pexy

SUMMARY:
The LIFT study will document the first clinical use of the ZiftLift Tissue Anchor in a browlift for patients with age-related brow ptosis. It is a single arm, open label multicenter study, to evaluate the safety and efficacy of the Zift Lift System. Up to 20 subjects in up to 3 sites will be enrolled in this study. Data from this trial will be used to confirm the device safety and efficacy and provide inputs to further refine the device design and procedure technique for future device iterations

DETAILED DESCRIPTION:
The LIFT study will document the first clinical use of the ZiftLift Tissue Anchor in a browlift for patients with age-related brow ptosis. It is a single arm, open label multicenter study, to evaluate the safety and efficacy of the Zift Lift System. Up to 20 subjects in up to 3 sites will be enrolled in this study. Data from this trial will be used to confirm the device safety and efficacy and provide inputs to further refine the device design and procedure technique for future device iterations Subjects with signed informed consents and who meet all the inclusion and none of the exclusion criteria and are treated with the device will be considered enrolled in the study. An interim report will be created after the first 20 patients has completed their 90 follow up and the data monitored. The 20 patients, 90 day report may be submitted to FDA and other agencies for product clearance and registrations. After FDA clearance has been obtained, the study may be converted to a post-market study for the long term follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to the treatment
2. Willing and able to participate in all the required follow-ups
3. Over 18 years of age
4. Under 75 years of age
5. Brow ptosis and/or functional limitations such as vision defects due to tissue laxity caused by aging

Exclusion Criteria:

1. Known allergies to local anesthesia
2. Currently undergoing chemotherapy or radiation therapy for cancer
3. Known advanced osteoporosis that may lead to skull thinning
4. Taking long-term immunosuppressant therapy
5. Taking chronic anticoagulation therapy (including ASA and NSAIDS) which can't be stopped for 10 days before treatment.
6. Unable or unwilling to participate in follow-up examinations
7. Evidence of brow soft tissue thickness less than 4mm by physical exam, ultrasound or direct probe (probe at the time of procedure)
8. Stroke or TIE (Transient Ischemic Event) within the past 6 months and currently on anti-platelet or other blood thinners
9. Chronic facial paralysis due to trauma, Bells Palsy, or similar etiology
10. Treatment with neurotoxin in the past 6 months and during the study period. Subjects may undergo a neurotoxin washout for 6 months prior to study participation
11. Planned surgical procedures, fillers or other facial procedures during the study period.
12. Planned modification of the eyebrows (to include plucking or shaving) during the study period
13. Planned MRI during the study period
14. Known nickel allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Brow Elevation | 90 days, 6 months, 1, 2, 3 and 4 years
  Change in brow elevation in mm from baseline to 90 days, with long term follow-up out to 4 years

SECONDARY OUTCOMES:
Patient Satisfaction | 90 days, 6 months, 1, 2, 3 and 4 years
  Patient Satisfaction using the Face-Q survey
Physician Satisfaction | 90 days, 6 months, 1, 2, 3 and 4 years
  Physician Satisfaction with Cosmetic Result. 7 metrics on all patients at all time points using a survey tool.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Hilger, MD, Principal Investigator — Centennial Lakes Surgery Center
Locations (1):
- Centennial Lakes Surgery Center, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No